CLINICAL TRIAL: NCT07110922
Title: Angiography and Electrogram Guided Bachmann Bundle Pacing - ANGEL BBP
Brief Title: Angiography and Electrogram Guided Bachmann Bundle Pacing
Acronym: (ANGEL-BBP)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pugazhendhi Vijayaraman (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Pugazhendhi Vijayaraman, Director, Cardiac Electrophysiology, Geisinger Clinic
Organization: Geisinger Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0403
Record Dates: First submitted 2025-06-24; First posted 2025-08-08 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases | interventions — Angiography; Electrocardiography

STUDY DESIGN:
Intervention Model Description: The study team will randomize 50 patients who satisfy inclusion and exclusion criteria to one of two arms - angiography only guided or angiography and ECG guided BBP lead implant. The study team will compare the difference in procedural success between the two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Angiography only (Experimental)
  Interventions: Diagnostic Test: Angiography only
- Angiography and ECG (Experimental)
  Interventions: Diagnostic Test: Angiography and ECG

INTERVENTIONS:
Diagnostic Test: Angiography only — Superior vena cava (SVC) angiogram will be used to anatomically identify the BB region
  Arms: Angiography only
Diagnostic Test: Angiography and ECG — Superior vena cava (SVC) angiogram will be used to anatomically identify the BB region and correlate with electrogram guidance for BBP
  Arms: Angiography and ECG

SUMMARY:
People eligible for this study are scheduled to have a permanent pacemaker (PPM) or defibrillator device (ICD) implanted as part of their routine care. This device will also have a wire placed in the right atrium (RA) of the heart. As an alternative to the RA, the wire can also be placed in the Bachmann bundle (BB).

This study is being done to compare two options to help place the wire in the Bachmann bundle. One option uses contrast dye and x-ray, and the other option uses electrocardiogram (ECG) and contrast dye and x-ray. We want to learn more about how well these options work in implanting the wire in the Bachmann bundle.

Both of these options are FDA approved and used in standard practice.

DETAILED DESCRIPTION:
The ANGEL BBP study is a prospective, single-center, randomized, controlled research study. The study team will identify all patients who satisfy the inclusion and exclusion criteria. The study team will evaluate the feasibility and success rates of Angiography guided Bachmann bundle pacing (BBP) lead implantation compared to traditional approach.

Eligible patients would undergo BBP using Medtronic 3830 lead and C304 or C315 family of sheaths. BBP will be confirmed at implant using Bachmann bundle potentials recorded from the lead, ECG 'P' wave morphology and duration during atrial pacing, fluoroscopic locations on right anterior oblique (RAO) and left anterior oblique (LAO) projections.

During implant procedure, 5-10 ml of contrast will be used to perform inferior superior vena cava (SVC) angiogram via the lead delivery sheath in RAO and LAO views. The pacing lead will be then implanted using these images as guidance along with recording of local electrograms from the pacing lead.

The study team will randomize 50 patients who satisfy inclusion and exclusion criteria. The study team will compare the difference in procedural success between Angiography and Electrogram guided BBP and Electrogram/ECG only guided BBP patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years of age
2. Patient with an indication for permanent pacemaker or ICD utilizing atrial pacing lead
3. Patient is willing to comply with all study procedures and be available for the duration of the study.

Exclusion Criteria:

1. Inability to provide informed consent
2. Pregnant
3. Enrolled in a concurrent study that may confound the results of this study.
4. Persistent atrial fibrillation at the time of implant (if cardioversion contraindicated at the time of implant, where BB mapping cannot be performed in sinus rhythm)
5. Renal dysfunction with serum Creatinine >3.0 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2027-09-26 (Estimated); Study Completion 2027-12-26 (Estimated)

PRIMARY OUTCOMES:
Success of Bachmann bundle pacing using angiography at implant | Perioperative
Change in implant procedure duration | Perioperative
  Change in implant procedure duration between the two arms

SECONDARY OUTCOMES:
Atrial pacing parameters | 3 month follow up
  atrial pacing parameters include threshold, sensing and impedance measured by device interrogation
Paced P-wave morphology compared to native P-waves | 3 month follow up
  P-wave morphology is measured via ECG at follow up and compared to native P-waves from baseline ECG
Paced P-wave duration compared to native P-waves | 3 month follow up
  P-wave duration is measured via ECG at follow up and compared to native P-waves from baseline ECG

CONTACTS AND LOCATIONS:
Overall Officials: Pugazhendhi Vijayaraman, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared in an identifiable way.